CLINICAL TRIAL: NCT02264015
Title: Pharmacodynamic Effects, Safety and Tolerability of 2 mg and 5 mg Cilobradine, Administered p.o. Once Daily Over 14 Days to Healthy Male and Female Volunteers in a Randomised, Placebo-controlled, Double Blind Study, With an Open-label Uncontrolled Intra-individual Comparison to 400 mg Moxifloxacin Single Dose in a Subset of Volunteers.
Brief Title: Pharmacodynamic Effects, Safety and Tolerability of Cilobradine, to Healthy Male and Female Volunteers, With an Intra-individual Comparison to Moxifloxacin in a Subset of Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 503.204
Record Dates: First submitted 2014-10-13; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — cilobradine; Moxifloxacin

ARMS (4):
- Cilobradine low (Experimental)
  Interventions: Drug: Cilobradine, low, film-coated tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo, film-coated tablets
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin, film-coated tablets
- Cilobradine high (Experimental)
  Interventions: Drug: Cilobradine, high, film-coated tablets

INTERVENTIONS:
Drug: Cilobradine, low, film-coated tablets
  Arms: Cilobradine low
Drug: Cilobradine, high, film-coated tablets
  Arms: Cilobradine high
Drug: Placebo, film-coated tablets
  Arms: Placebo
Drug: Moxifloxacin, film-coated tablets
  Arms: Moxifloxacin

SUMMARY:
Incidence of visual phenomena, heart rate at rest, safety (with particular emphasis on QT analysis of ECGs), and pharmacokinetic parameters

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), clinical laboratory tests

   1.1 No finding deviating from normal and of clinical relevance

   1.2 No evidence of a clinically relevant concomitant disease
2. Age ≥21 and Age ≤55 years
3. BMI ≥18.5 and BMI < 30 kg/m2 (Body Mass Index)
4. Resting Heart rate (HR) (after 10 min. in the supine position) of equal or more than 60 bpm
5. Females: post-menopausal or those who have had a hysterectomy (plus a negative pregnancy test)
6. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, ophthalmological, or hormonal disorders
2. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
3. History of relevant orthostatic hypotension, fainting spells or blackouts
4. Chronic or relevant acute infections
5. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
6. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
7. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
8. Participation in another trial with an investigational drug within two months prior to administration or during the trial
9. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes/day)
10. Inability to refrain from smoking on trial days
11. Alcohol abuse
12. Drug abuse
13. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
14. Excessive physical activities (within one week prior to administration or during the trial)
15. Any laboratory value outside the reference range that is of clinical relevance.

    Exclusion criteria specific for this study:
16. Subjects at increased risk for development of cardiac arrhythmia (e.g. family history of long QT syndrome or sudden cardiac death)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2004-01; Primary Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Incidence of visual phenomena | Up to 12 days after last scheduled study day
  Reported as adverse events
Change in heart rate at rest | Pre dose, up to 12 hours after drug administration

SECONDARY OUTCOMES:
Investigator assessed tolerability on a 4 point scale | Up to 12 days after last scheduled study day
Number of participants with abnormal findings in physical examination | Up to 12 days after last scheduled study day
Number of participants with clinically significant changes in vital signs | Up to 12 days after last scheduled study day
Number of participants with adverse events | Up to 12 days after last scheduled study day
Characteristics of visual phenomena on a special questionnaire | Up to 12 days after last scheduled study day
Number of participants with abnormal changes in clinical laboratory parameters | Up to 12 days after last scheduled study day
Number of participants with abnormal findings in electrocardiogram (ECG) | Up to 12 days after last scheduled study day
Area under the concentration-time curve of the analyte in plasma from zero time to 24 hours (AUC0-24) | Up to 24 hours after drug administration
Maximum plasma concentration following the first dose (Cmax) | Up to 24 hours after drug administration
Time from first dose to the maximum plasma concentration (tmax) | Up to 24 hours after drug administration
Terminal half-life (t1/2) | Up to 24 hours after drug administration
Mean residence time of the analyte in the body after oral administration (MRTpo) | Up to 24 hours after drug administration
Apparent clearance of the analyte in plasma following extravascular administration (CL/F) | Up to 24 hours after drug administration
Apparent volume of distribution during the terminal phase λz following extravascular administration (Vz/F) | Up to 24 hours after drug administration